CLINICAL TRIAL: NCT00650806
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Investigate the Safety and Efficacy of JNJ-28431754 in Nondiabetic Overweight and Obese Subjects
Brief Title: A Study of the Safety and Effectiveness of Canagliflozin (JNJ-28431754) in Promoting Weight Loss in Overweight and Obese Patients Who do Not Have Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014578; 28431754OBE2001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Weight loss; Anti-Obesity Agents; Human
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Canagliflozin 50 mg (Experimental): Each patient will receive 50 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Canagliflozin 300 mg (Experimental): Each patient will receive 300 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Placebo (Placebo Comparator): Each patient will receive matching placebo once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) — One 50 mg, 100 mg, or 300 mg over-encapsulated tablet orally (by mouth) once daily for 12 weeks.
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg; Canagliflozin 50 mg
Drug: Placebo — One matching placebo capsule orally once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and effectiveness of JNJ-28431754 in promoting weight loss in patients who are overweight or obese and who do not have diabetes.

DETAILED DESCRIPTION:
The prevalence of obesity is increasing worldwide. Obesity and being overweight are major risk factors for chronic cardiovascular disease, type 2 diabetes mellitus, hypertension and stroke, and certain types of cancers. JNJ-28431754 is being investigated in this study for its possible effectiveness in promoting weight loss when taken over a 12-week period. The study consists of 3 phases: a pretreatment phase that includes a 7-day screening period and a 4-week run-in period, a 12-week double-blind treatment phase (neither the patient nor the investigator will know which treatment the patient is receiving) with an end-of-treatment visit, and a posttreatment phase. In the pretreatment phase, after giving written informed consent, patients will undergo screening evaluations. Patients who successfully complete the screening period will enter the 4-week run-in period and be given dietary and exercise counseling as standardized non-drug therapy for weight loss. During the 12 weeks of treatment, all patients will continue on the study diet and exercise non-drug therapy and will visit the study site about every 3 weeks to have their weight and the results of other safety and effectiveness tests recorded, and to have blood samples collected to measure the concentration of JNJ-28431754 in their blood. In the posttreatment phase, patients will return to the study site for a follow-up visit 14 days after receiving their last dose of study drug. Patient safety will be monitored throughout the study using spontaneous adverse event reporting, clinical laboratory tests (hematology, serum chemistry, urinalysis); pregnancy tests; physical examinations; electrocardiograms; vital signs measurements; overnight urine collection to measure albumin excretion; assessment of calcium and phosphate homeostasis (balance), bone formation and reabsorption markers, and hormones regulating calcium and phosphorus homeostasis; and self administered vaginal and urine sample collection for fungal and bacterial culture in subjects with symptoms consistent with vulvovaginal candidiasis and urinary tract infection. Patients will complete 2 questionnaires to record their reactions to taking the study drug and the effect of body weight on their daily lives. About 100 patients of the approximately 400 who qualify for the study, and who consent to this, will take part in 2 oral glucose tolerance tests (OGTTs). During the OGTTs they will drink a glucose solution and have a series of blood samples collected to measure glucose concentration, collect their urine over a 2 hour period, and (at the second OGTT only) have blood samples collected to measure JNJ 28431754 blood concentrations. The primary clinical theory for this study is that at well-tolerated doses, JNJ-28431754 is superior to placebo as measured by the percent change in body weight from baseline (Day 1 of the double-blind treatment period) through Week 12.

ELIGIBILITY:
Inclusion Criteria:

* BMI >=30 kg/m2 and <50 kg/m2 or a BMI >=27 kg/m2 and <50 kg/m2 in the presence of controlled hypertension and/or treated or untreated dyslipidemia
* Must have a stable weight, i.e., increasing or decreasing not more than 5% in the 3 months before screening
* Serum creatinine <=1.5 mg/dL for men and <=1.4 mg/dL for women at screening
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels within 2 times the upper limit of normal (ULN) and bilirubin within the normal range, unless the findings are consistent with Gilbert's disease
* fasting plasma glucose PG <7.0 mmol/L (126 mg/dL) at screening

Exclusion Criteria:

* A history of hereditary glucose-galactose malabsorption or primary renal glycosuria
* An established diagnosis of diabetes mellitus or treatment with glucose lowering drugs at screening
* A history of reactive hypoglycemia or of symptomatology possibly due to hypoglycemia
* Fasting triglyceride level >6.78 mmol/L (600 mg/dL) at screening
* History of obesity with a known cause (e.g., Cushing's disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (36):
- United States (35):
  - Hot Springs, Arkansas
  - Walnut Creek, California
  - Westlake Village, California
  - Destin, Florida
  - Jacksonville, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Stockbridge, Georgia
  - Boise, Idaho
  - Eagle, Idaho
  - Meridian, Idaho
  - Evansville, Indiana
  - Overland Park, Kansas
  - Witchita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Auburn, Maine
  - Milford, Massachusetts
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Manilus, New York
  - Medford, Oregon
  - Portland, Oregon
  - Goose Creek, South Carolina
  - Mt. Pleasant, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Dallas, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - West Jordan, Utah
  - Norfolk, Virginia
  - Wauwatosa, Wisconsin
- Ponce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin (JNJ-28431754) in nondiabetic, overweight, and obese patients. The study was conducted between 31 March 2008 and 18 September 2008 and recruited patients from 38 study centers located in the United States and Puerto Rico.
Pre-assignment Details: A total of 376 patients were randomly allocated to the 4 treatment arms in the study and comprised the intent-to-treat analysis set which was used for the efficacy analyses. All 376 patients received at least 1 dose of study drug and were included in the safety analysis set.
Groups:
- Placebo: Each patient received matching placebo once daily for 12 weeks.
- Canagliflozin 50 mg: Each patient received 50 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
- Canagliflozin 300 mg: Each patient received 300 mg of canaliflozin (JNJ-28431754) once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 89 | 98 | 93 | 96
Completed | 71 | 77 | 64 | 70
Not Completed | 18 | 21 | 29 | 26
Not completed — Adverse Event | 0 | 5 | 3 | 4
Not completed — Lost to Follow-up | 7 | 6 | 11 | 10
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 5 | 8 | 6
Not completed — Noncompliance with study drug regimen | 1 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 2 | 3 | 5 | 4
Not completed — Other | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 89 | 98 | 93 | 96 | 376
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 88 | 97 | 93 | 94 | 372
  >=65 years | 1 | 1 | 0 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 45.1 (11.92) | 44.9 (11.8) | 45.8 (10.95) | 43.5 (10.99) | 44.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 86 | 76 | 86 | 323
  Male | 14 | 12 | 17 | 10 | 53
Region Enroll [Number; unit: participants]
  PUERTO RICO | 3 | 4 | 4 | 5 | 16
  UNITED STATES | 86 | 94 | 89 | 91 | 360

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight From Baseline to Week 12
Description: The table below shows the mean percent change in body weight from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the least-squares mean percent change.
Time Frame: Day 1 (Baseline) and Week 12
Population: This analysis was conducted using the intent-to-treat analysis set, which included all patients who were randomly assigned to a treatment group. The last-observation-carried-forward method was applied when the Week 12 values were missing. The table includes only patients with both baseline and post baseline values.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Canaglifloziin 300 mg: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canaglifloziin 300 mg
Number analyzed (Participants) | 86 | 95 | 85 | 93
Percent change | -1.1 (2.4) | -2.0 (3.0) | -2.8 (2.9) | -2.5 (3.0)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg; Test type: Superiority or Other; p = 0.031, ANOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center; Least-Squares Mean Difference = -0.9, 95% CI 2-sided [-1.6 to -0.1], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center; Least-Squares Mean Difference = -1.6, 95% CI 2-sided [-2.4 to -0.8], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Placebo vs Canaglifloziin 300 mg; Test type: Superiority or Other; p < 0.001, ANOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center; Least-Squares Mean Difference = -1.4, 95% CI 2-sided [-2.1 to -0.6], Standard Error of Mean 0.4

2. Secondary Outcome: Absolute Change in Body Weight From Baseline to Week 12
Description: The table below shows the mean absolute change in body weight from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 86 | 95 | 85 | 93
kg | -1.1 (2.46) | -1.9 (2.90) | -2.8 (2.90) | -2.4 (2.90)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg; Test type: Superiority or Other; p = 0.045, ANCOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center. Baseline body weight was a covariate; Least-Squares Mean Difference = -0.8, 95% CI 2-sided [-1.58 to -0.02], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center. Baseline body weight was a covariate; Least-Squares Mean Difference = -1.6, 95% CI 2-sided [-2.40 to -0.80], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.001, ANCOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center. Baseline body weight was a covariate; Least-Squares Mean Difference = -1.3, 95% CI 2-sided [-2.07 to -0.51], Standard Error of Mean 0.40

3. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline to Week 12
Description: The table below shows the mean change in BMI from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 86 | 95 | 85 | 93
kg/m2 | -0.4 (0.86) | -0.7 (1.05) | -1.0 (1.05) | -0.9 (1.07)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg; Test type: Superiority or Other; p = 0.031, ANCOVA; Cofactors were treatment, run-in weight loss stratum, and pooled center. The corresponding baseline measurement was a covariate; Least-Squares Mean Difference = -0.31, 95% CI 2-sided [-0.59 to -0.03], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -0.6, 95% CI 2-sided [-0.90 to -0.32], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -0.48, 95% CI 2-sided [-0.76 to -0.20], Standard Error of Mean 0.14

4. Secondary Outcome: Percentage of Patients Who Lost at Least 5% of Their Initial Body Weight by Week 12
Description: The table below shows the percentage of patients who lost at least 5% of their initial body weight by Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo).
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 86 | 95 | 85 | 93
Percentage of patients | 8.1 | 12.6 | 18.8 | 17.2
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel — P-value controlled for run-in weight loss stratum and pooled center; Odds Ratio (OR) = 1.7, 95% CI [0.6 to 5.6] — Odds ratio and Confidence Interval controlled for run-in weight loss stratum and pooled center
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.059, Cochran-Mantel-Haenszel — P-value controlled for run-in weight loss stratum and pooled center; Odds Ratio (OR) = 2.9, 95% CI 2-sided [0.9 to 11.1] — Odds ratio and Confidence Interval controlled for run-in weight loss stratum and pooled center
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.027, Cochran-Mantel-Haenszel — P-value controlled for run-in weight loss stratum and pooled center; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.0 to 10.0] — Odds ratio and Confidence Interval controlled for run-in weight loss stratum and pooled center

5. Secondary Outcome: Percentage of Patients Who Lost at Least 10% of Their Initial Body Weight by Week 12
Description: The table below shows the percentage of patients who lost at least 10% of their initial body weight by Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo).
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 86 | 95 | 85 | 93
Percentage of patients | 0.0 | 3.2 | 2.4 | 1.1
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg; Test type: Superiority or Other; p = 0.117, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test controlled for run-in weight loss stratum and pooled center
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.225, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test controlled for run-in weight loss stratum and pooled center
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test controlled for run-in weight loss stratum and pooled center

6. Secondary Outcome: Change in Waist Circumference From Baseline to Week 12
Description: The table below shows the mean change in waist circumference from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 78 | 87 | 73 | 82
cm | -1.2 (10.06) | -1.4 (4.99) | -2.9 (10.32) | -2.6 (7.22)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg; Test type: Superiority or Other; p = 0.835, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -0.26, 95% CI 2-sided [-2.68 to 2.17], Standard Error of Mean 1.23
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.466, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -0.94, 95% CI 2-sided [-3.47 to 1.59], Standard Error of Mean 1.29
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.273, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Sqaures Mean Difference = -1.37, 95% CI 2-sided [-3.87 to 1.09], Standard Error of Mean 1.25

7. Secondary Outcome: Change in Hip Circumference From Baseline to Week 12
Description: The table below shows the mean change in hip circumference from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Canaglifozin 50 mg: Each patient received 50 mg of canagliflozin (JNJ-28431754) once daily for 12 weeks.
Arm/Group | Placebo | Canaglifozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 77 | 86 | 72 | 81
cm | 0.1 (10.38) | -2.0 (3.97) | -2.1 (10.62) | -3.0 (7.95)
Statistical Analysis 1: Comparison: Placebo vs Canaglifozin 50 mg; Test type: Superiority or Other; p = 0.149, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -1.63, 95% CI 2-sided [-3.85 to 0.59], Standard Error of Mean 1.13
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.541, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -0.72, 95% CI 2-sided [-3.05 to 1.6], Standard Error of Mean 1.18
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.121, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = -1.78, 95% CI 2-sided [-4.03 to 0.47], Standard Error of Mean 1.15

8. Secondary Outcome: Change in Waist/Hip Ratio From Baseline to Week 12
Description: The table below shows the mean change in waist/hip ratio from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Canaglifozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 77 | 86 | 72 | 81
ratio | -0.011 (0.0542) | 0.003 (0.0422) | -0.008 (0.0915) | -0.004 (0.0469)
Statistical Analysis 1: Comparison: Placebo vs Canaglifozin 50 mg; Test type: Superiority or Other; p = 0.239, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = 0.011, 95% CI 2-sided [-0.0071 to 0.0286], Standard Error of Mean 0.0091
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority or Other; p = 0.900, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = 0.001, 95% CI 2-sided [-0.0174 to 0.0198], Standard Error of Mean 0.0095
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 300 mg; Test type: Superiority or Other; p = 0.822, ANCOVA; [statistical method as in outcome 3, analysis 1]; Least-Squares Mean Difference = 0.002, 95% CI 2-sided [-0.0160 to 0.0202], Standard Error of Mean 0.0092

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 12 weeks.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Arm/Group | Placebo | Canagliflozin 50 mg | Canagliflozin 100 mg | Canagliflozin 300 mg
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/98 | 0/93 | 0/96
Other Adverse Events (participants affected / at risk) | 28/89 | 41/98 | 30/93 | 31/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=89) | Canagliflozin 50 mg (N=98) | Canagliflozin 100 mg (N=93) | Canagliflozin 300 mg (N=96)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=89) | Canagliflozin 50 mg (N=98) | Canagliflozin 100 mg (N=93) | Canagliflozin 300 mg (N=96)
Constipation (Gastrointestinal disorders) | 2 | 5 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 7 | 6 | 3
Nasopharyngitis (Infections and infestations) | 3 | 6 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 6 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 6 | 5
Urinary tract infection (Infections and infestations) | 6 | 10 | 7 | 8
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 8 | 5 | 14
Headache (Nervous system disorders) | 7 | 6 | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.